CLINICAL TRIAL: NCT05654740
Title: Design of the Virtual Leisure Pilot Study - Virtual Reality Delivered Stress Reduction, Entertainment, and Distraction at a Closed Psychiatric Ward
Brief Title: Virtual Leisure - Virtual Reality Delivered Recreation at a Closed Psychiatric Ward
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1000
Record Dates: First submitted 2022-11-08; First posted 2022-12-16 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2022-12

CONDITIONS: Psychiatric Hospitalization
Keywords: Psychiatric in-patient care; Virtual Reality; Coercion; Stress reduction; Entertainment; Distraction

STUDY DESIGN:
Intervention Model Description: We will compare outcomes for a 12-month period where all patients are offered Virtual Reality experiences regularly to outcomes for a 12-month period with no availability of Virtual Reality experiences in one specified closed psychiatric ward.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality experiences (Experimental): Virtual Reality experiences are offered regularly
  Interventions: Device: Virtual Reality Experiences
- No Virtual Reality (No Intervention): Virtual Reality experiences are not offered

INTERVENTIONS:
Device: Virtual Reality Experiences — Virtual Reality experiences including stress reduction, distraction and entertainment
  Arms: Virtual Reality experiences

SUMMARY:
Background: The environment at a psychiatric in-patient ward can lead to emotional distress and behavioral deviations in vulnerable individuals potentially resulting in conflicts, increased use of need-based medication and coercive actions, along with low satisfaction with treatment. To accommodate these challenges recreational and entertaining interventions are generally recommended. The tested interventions have, however, shown varying effects and often demand a high degree of planning and staff involvement while also being difficult to adapt to individual needs. Virtual Reality (VR) may help overcome these challenges.

Methods: The study is a clinical trial, employing a mixed-methods design, enrolling 124 patients hospitalized at one closed psychiatric ward in the capital region of Denmark. All patients will be offered VR based stress reduction (e.g., mindfulness/relaxation techniques), entertainment, and distraction regularly during their hospitalization. Feasibility and acceptability will be explored with qualitative interviews supplemented with repeated non-participants observations and focus groups. The effect of the intervention will be assessed by comparing quantitative outcomes (e.g., coercion, need-based medication, and perceived stress) for a 12-month period with VR experiences available to a 12-month period without VR experiences available.

Discussion: It is of significant interest to find non-intrusive interventions with minimal side-effects that may provide an alternative to pharmacological interventions and coercive actions in mental health services. If the VR intervention is found to be feasible and acceptable a larger study can be initiated and if found to be effective in a psychiatric in-patient setting, it can be scaled for use in psychiatric treatment facilities in general where it may benefit a large group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a closed psychiatric ward
* Ability to give informed consent

Exclusion Criteria:

* Significantly impaired vision hindering engagement in Virtual Reality experiences

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability | up to 26 weeks
  ≥80% of the in-patients' consent to participating in the study

SECONDARY OUTCOMES:
Need-based medication | up to 26 weeks
  Use of need-based medication (e.g. benzodiazepines and antipsychotic medication)
Client Satisfaction | up to 26 weeks
  The Client Satisfaction Questionnaire will be used to assess patients satisfaction with treatment.
Coercive actions | up to 26 weeks
  Coercive actions during patient's hospitalization and the closed psychiatric ward. Coercive actions comprise mechanical restraint (belt fixation) and forced sedation (injecting the patient with sedating medication without their consent to diminish aggressive behavior)

OTHER OUTCOMES:
Global perceived level of stress over the past week | up to 26 weeks
  Measured by the Perceived Stress Scale, assessing the degree to which situations are appraised as stressful.
Distress before and after using Virtual Reality | up to 26 weeks
  Measured by the Subjective Units of Distress Scale (SUDS) which measures the intensity of feelings and other internal experiences, such as anxiety, anger, agitation, stress or other painful feelings.
Number of days hospitalized. | up to 26 weeks
Risk of violence within the next 24 hours | up to 26 weeks
  Measured three times a day with the Brøset Violence Checklist (BVC) as part of standard procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Clemmensen, PhD, Principal Investigator — Psykiatrisk Center København
Locations (1):
- Mental Health Centre Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clemmensen L, Jorgensen G, Gundersen KB, Smith LC, Midtgaard J, Bouchard S, Thomsen CP, Turgut L, Glenthoj LB. Study protocol for virtual leisure investigating the effect of virtual reality-delivered stress reduction, entertainment and distraction on the use of coercion and need-based medication and patient satisfaction at a closed psychiatric intensive care unit - a mixed-methods pilot clinical trial. BMJ Open. 2023 Sep 22;13(9):e070566. doi: 10.1136/bmjopen-2022-070566. PMID 37739476